CLINICAL TRIAL: NCT04886609
Title: ORISE Study: Evaluation of Novel Injecting Solution (ORISE) During Endoscopic Resection of Colorectal Polyps.
Acronym: ORISE
Status: Terminated | Type: Observational
Why Stopped: Safety issues/concerns with device use reported by the manufacturer and requested product recall and to stop use of product.
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 275810
Record Dates: First submitted 2021-05-10; First posted 2021-05-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Colorectal Polyp
Keywords: ORISE gel; EMR; ESD; Colorectal polyps; submucosal injection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: ORISE gel — To establish if ORISE Gel an effective and feasible submucosal injecting solution during endoscopic resection of large colorectal polyps

SUMMARY:
Is ORISE Gel an effective and feasible submucosal injecting solution during endoscopic resection of large colorectal polyps.

DETAILED DESCRIPTION:
Endoscopic resection of large colonic polyps is preferred over Surgical resections due to lower morbidity and preservation of the colon and its functions.

The use of submucosal injection is essential for a successful resection (EMR/ ESD). Injection of fluid into the submucosa cushions and isolates the tissue just before capture of the target lesion with a snare, thereby reducing thermal injury and the risk of perforation during EMR. ESD requires a long period of submucosal dissection and that involves multiple injections to maintain the submucosal cushion; without which the risk of perforation increases.

A mixture of normal saline solution + epinephrine and blue dye like indigo carmine is the commonly used injecting solution. However, Saline dissipates very quickly leading to frequent and multiple injections. This leads to longer procedure time.

Studies have demonstrated long-lasting effects of colloids when injected in the submucosal space. ORISE gel is a newly licensed injecting solution which contains a poloxamer agent leading to longer lasting submucosal cushion effect.

Multicentre prospective observational cohort study

Primary Objective : Primary Objective To evaluate the technical feasibility, effectiveness & safety of the ORISE gel as an injecting solution on its own during endoscopic resection of colorectal polyps (ability to start and finish the resection with ORISE).

Secondary Objective : To identify Polyp Resection Time (PRT) and the amount of ORISE gel used during resection of large colorectal polyps.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old at the date of consent
* Subjects referred for EMR for the excision of:

Treatment naïve, laterally spreading sessile, flat polyps or adenomas of the colon equal to or greater than 20 mm in largest dimension, assessed by the investigator to be suitable for EMR or ESD.

Exclusion Criteria:

* Lesions less than 20 mm in largest dimension
* Subjects with ulcerated depressed lesions (Paris type III-excavated) or biopsy proven invasive carcinoma
* Scarred polyps
* Endoscopic appearance of deep invasive malignancy
* Previous partial resection or attempted resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients undergoing EMR or ESD at each recruiting centre who meet below eligibility criteria will be invited to participate.
Sampling Method: Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2023-01-12 (Actual); Study Completion 2023-01-12 (Actual)

PRIMARY OUTCOMES:
Feasability | 1 year
  Ease of use, rated on a 5-point visual analog scale for: very easy, easy, neutral, difficult and very difficult.
Effectiveness | 1 year
  Number of patients where alternatives to ORISE gel had to be used to complete the procedure
Safety - Presence of Muscle fibers in the resected specimen | 1 year
  Presence of Muscle fibers in the resected specimen
Safety - Complications | 1 year
  Complications: Perforationpost polypectomy syndrome, Intra procedural bleeding, post procedural

SECONDARY OUTCOMES:
Total injected volume per lesion size | 1 year
  Total injected volume per lesion size: calculated by dividing the injected volume needed to complete the EMR procedure (in mL) by the lesion size (in mm2).
Sydney Resection Quotient | 1 year
  Sydney Resection Quotient: calculated by dividing the lesion size (in mm2) by the number of resections required to remove the lesion
Feasability | 1 year
  Polyp Resection Time

CONTACTS AND LOCATIONS:
Overall Officials: Pradeep Bhandari, Prof, Principal Investigator — Portsmouth Hospitals University NHS Trust
Locations (5):
- Humaitas Research Hospital, Milan, Italy
- United Kingdom (4):
  - Portsmouth Hospital NHS Trust, Portsmouth, Hampshire
  - Leeds General Infirmary, Leeds
  - Kings College Hospital, London
  - John Radcliffe Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Undecided
Non identifiable Data regards primary and secondary outcome measures to be shared with other investigators